CLINICAL TRIAL: NCT06694610
Title: A Study on the Relationship Between Individualized Low Voltage Regions in Left Atrium and the Mechanism of Atrial Fibrillation in Persistent Atrial Fibrillation Under Ultra-High-Resolution Mapping
Acronym: ILVRA-PAFM-UAH
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Third People's Hospital of Chengdu (Other)
Responsible Party: Principal Investigator, Hanxiong Liu, Principal Investigator, The Third People's Hospital of Chengdu
Allocation: Not Applicable | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CDSY-ILVRA-PAFM-UAH
Record Dates: First submitted 2024-11-12; First posted 2024-11-19 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-11

CONDITIONS: Atrial Fibrillation Recurrent
Keywords: 心房颤动（Atrial Fibrillation）

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- non-pulmonary vein ablation group (Experimental): In the non-pulmonary vein ablation group, pulmonary vein isolation was not allowed, but the left atrial low-voltage area was treated first, and then the ablation route that terminated the reentry ring was treated.
  Interventions: Procedure: non-pulmonary vein ablation group
- only pulmonary vein ablation group (Active Comparator): In the group treated with only pulmonary vein ablation route, only potential isolation of pulmonary vein was performed, and bidirectional block was the end point.
  Interventions: Procedure: only pulmonary vein ablation group

INTERVENTIONS:
Procedure: non-pulmonary vein ablation group — In the non-pulmonary vein ablation group, pulmonary vein isolation was not allowed, but the left atrial low-voltage area was treated first, and then the ablation route that terminated the reentry ring was treated.
  Arms: non-pulmonary vein ablation group
Procedure: only pulmonary vein ablation group — In the group treated with only pulmonary vein ablation route, only potential isolation of pulmonary vein was performed, and bidirectional block was the end point.
  Arms: only pulmonary vein ablation group

SUMMARY:
The latest OCTARAY multi-electrode mapping catheter and TUREref technology were used to perform ultra-high precision mapping on the left atrial and left atrial auricle of persistent atrial fibrillation in the condition of sinus rhythm and atrial fibrillation respectively, and the density and accuracy of potential were significantly improved. According to the mapping results, the numerical calculation of the personalized low voltage region was carried out, and the personalized ablation route was designed according to the low voltage region.

DETAILED DESCRIPTION:
1. The latest OCTARAY multi-electrode mapping catheter and TUREref technology were used to perform ultra-high precision mapping on the left atrial and left atrial auricle of persistent atrial fibrillation in the condition of sinus rhythm and atrial fibrillation respectively, and the density and accuracy of potential were significantly improved. According to the mapping results, the numerical calculation of the personalized low voltage region was carried out, and the personalized ablation route was designed according to the low voltage region.
2. Octaray multi-electrode mapping catheter and CartoFinder software were used to map focal drive and reentrant ring in left atrial fibrillation. Based on the CartoFinder software's mapping of focal drive and normal potential areas, potential analysis was used to find the reentrant ring of persistent AF. The ablation route of the reentry ring is designed.
3. Based on the designed ablation route, it is divided into different ablation route groups. They were divided into two groups: treatment of pulmonary vein ablation route only; Treatment of non-pulmonary venous ablation route group. In the group treated with only pulmonary vein ablation route, only potential isolation of pulmonary vein was performed, and bidirectional block was the end point. In the non-pulmonary vein ablation group, pulmonary vein isolation was not allowed, but the left atrial low-voltage area was treated first, and then the ablation route that terminated the reentry ring was treated. In the low-voltage region ablation group, if there was a large difference between the low-voltage region in atrial fibrillation and the low-voltage region in sinusional state, there was a common low-voltage region and a non-common low-voltage region. The non-common low-voltage region refers to the region with low voltage region in atrial fibrillation and no low voltage region in sinusional state. This type of cases were divided into two subgroups, A and B. Group A preferentially ablated the non-common low voltage region, group B preferentially ablated the common low voltage region. In the condition of atrial fibrillation, if there is overlap between the low-voltage ablation line and the reentrant ablation line in the non-pulmonary vein ablation group, the overlap line should be abated preferentially.
4. In each group, the atrial fibrillation was attributed to the maintenance factor group according to the region of transsinus ablation or the region of atrial flutter tachycardia ablation. Pulmonary vene-associated atrial fibrillation, low-voltage region associated atrial fibrillation, reentrant ring associated atrial fibrillation.
5. The intraoperative ablation data of each group were analyzed, such as ablation number, time, stopping site, and follow-up sinus rhythm maintenance rate. "Follow-up times are at 3 months, 6 months, and 12 months post-surgery. "Monitoring heart rhythm through the use of 7-day ambulatory Holter monitoring."

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 18 to 85 years;
2. Diagnosed with drug-refractory, symptomatic, persistent atrial fibrillation; Definition: At least one electrocardiogram (ECG) record of an atrial fibrillation episode within 12 months prior to enrollment.
3. Non-valvular atrial fibrillation;
4. Able to understand the purpose of the study, voluntarily participate in the study, the patient or their legal representative signs the informed consent form, and willing to complete follow-ups as required by the study protocol.-

Exclusion Criteria:

1. Atrial fibrillation secondary to thyroid disease or other reversible factors;
2. Imaging studies indicating intracardiac thrombus;
3. Moderate to severe mitral stenosis or regurgitation;
4. Left ventricular ejection fraction <40%, or New York Heart Association (NYHA) functional class III or IV;
5. Unstable angina;
6. Myocardial infarction (MI) or coronary artery bypass grafting (CABG) within 3 months prior to enrollment;
7. Presence of mural thrombus, space-occupying disease, or other abnormalities that hinder vascular puncture or catheter manipulation;
8. Contraindications to anticoagulation and a history of blood coagulation or bleeding abnormalities;
9. Patients with active systemic infections; Patients who have had an atrial septal closure device implanted within the last 6 weeks;
10. Female patients who are pregnant, breastfeeding, or unable to use contraception during the study period;
11. Patients with a life expectancy of less than 12 months (e.g., advanced malignant tumors); patients who have had an atrial septal closure device implanted within the last 6 weeks;
12. Conditions affecting vascular access;
13. Patients who are concurrently participating in other drug or device clinical trials;
14. Any other abnormalities or diseases that the investigator deems should exclude the patient from the study enrollment.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-11-15 (Estimated); Primary Completion 2025-04-05 (Estimated); Study Completion 2026-04-05 (Estimated)

PRIMARY OUTCOMES:
Immediate Atrial Fibrillation Termination Rate | Intraoperative Immediate
  The number of atrial fibrillation rhythms ablated to sinus rhythm or flutter/atrial tachycardia during the procedure.

SECONDARY OUTCOMES:
Ablation Success Rate at 12 Months Post-Operation. | 12 Months Post-Operation.
  No electrocardiogram (ECG) recordings of atrial fibrillation, flutter, or tachycardia lasting ≥30 seconds from the end of the blanking period to the end of the 12-month follow-up.

OTHER OUTCOMES:
The number and location of re-entrant circuits mapped during surgery | Intraoperative Immediate
the location of ablation to sinus rhythm or flutter | Intraoperative Immediate
the number of three-dimensional mapping points | Intraoperative Immediate

IPD SHARING:
Plan to Share IPD: Undecided